CLINICAL TRIAL: NCT04475380
Title: Complex All-comers and Patients With Diabetes or Prediabetes, Treated With Xience Sierra Everolimus-eluting Stents (COASTLINE)
Brief Title: Complex All-comers and Patients With Diabetes or Prediabetes, Treated With Xience Sierra Everolimus-eluting Stents
Status: Completed | Type: Observational
Sponsor: Foundation of Cardiovascular Research and Education Enschede (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: COASTLINE
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis
Keywords: Drug-eluting stent; Durable polymer; Everolimus; All comers population; High-risk all comers; Target vessel failure; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Angina, Unstable; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All-comer patients requiring PCI: All-comer patients requiring percutaneous coronary intervention (PCI) for the treatment of significant coronary artery of bypass graft lesions that are suitable for treatment with Xience Sierra DES
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI for treatment of coronary or bypass graft lesions

SUMMARY:
Drug eluting stents (DES) are widely used for treatment of coronary artery lesions. The Xience Sierra stent has a refined design of the metal stent backbone and is used in patients with various clinical syndromes and in different lesions. Clinical outcome of patients with previously unknown (silent) diabetes and prediabetes is of increasing interest since the latter group has recently shown to be associated with a significant risk of adverse cardiovascular events after treatment with contemporary DES. Outcome data in a population of high-risk all-comer patients, including many patients with diabetes mellitus and prediabetes, would be of great interest, but such data are not available yet. In addition, there is a lack of data in a general all-comer population. Therefore, the COASTLINE study will primarily assess the safety and efficacy of the Xience Sierra stent in a general all-comer population as well as a high-risk all-comer population.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* requiring PCI and treated with Xience Sierra
* capable of providing informed consent

Exclusion Criteria:

* known intolerance to components of the study DES or antithrombotic/anticoagulant therapy
* planned elective surgery necessitating interruption of dual antiplatelet therapy (DAPT) < 3 months
* patient is known to be pregnant, unlikely to adhere to follow-up or expected live < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers. Patients for elective PCI or acute PCI
Sampling Method: Probability Sample
Enrollment: 1757 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Target vessel failure (TVF) at 1-year follow up in complex all-comers | 1 year
  TVF is a composite endpoint consisting of cardiac death, target vessel related myocardial infarction, or clinically driven target vessel revascularization.
Target lesion failure (TLF) at 2-year follow up in all-comers | 2 year
  TLF is a composite endpoint consisting of cardiac death, target vessel related myocardial infarction, or clinically driven target lesion revascularization.

SECONDARY OUTCOMES:
TVF at 2 year follow up | 2 year
Death | up to 3 year
  any/cardiac/non-cardiac
Myocardial infarction | up to 3 year
  target vessel related/any/periprocedural
Clinically indicated target vessel revascularization | up to 3 year
Clinically indicated target lesion revascularization | up to 3 year

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Thoraxcentrum Twente, Enschede
  - Haga Ziekenhuis, The Hague

REFERENCES:
- [Derived] van Vliet D, Ploumen EH, Pinxterhuis TH, Buiten RA, Aminian A, Schotborgh CE, Anthonio RL, Zocca P, Hartmann M, Stoel MG, de Man FHAF, Linssen GCM, Doggen CJM, van der Heijden LC, Kok MM, von Birgelen C. Complex all-comers and patients with diabetes and prediabetes treated with Xience Sierra everolimus-eluting stents: COASTLINE high-risk. Eur Heart J Open. 2025 Oct 21;5(6):oeaf140. doi: 10.1093/ehjopen/oeaf140. eCollection 2025 Nov. PMID 41230396